CLINICAL TRIAL: NCT06758609
Title: Local Hypothermia and Endovascular Recanalization for Acute Large Artery Occlusive Stroke-A Multicenter, Prospective, Open-label, Blinded-Endpoint, Randomized Controlled Trial
Brief Title: To Assess the Effectiveness and Safety of Catheter-based Focal Intracranial Hypothermia Combined with Endovascular Reperfusion Therapy for Patients with Acute Anterior Circulation Large Artery Occlusion
Acronym: CHILL-ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Zhixin Huang, Principal Investigator, Guangdong Second Provincial General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHILL-ART
Record Dates: First submitted 2024-12-20; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Acute Cerebrovascular Accident; Acute Ischemic Stroke; Internal Carotid Artery; Middle Cerebral Artery Occlusion
MeSH Terms: conditions — Stroke; Ischemic Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanical thrombectomy combined with intra-arterial selective cooling infusion (hypothermia) group (Experimental): Patients received a total of 350 ml of 4°C saline infusion in addition to mechanical thrombectomy (MT).
  Interventions: Procedure: Mechanical thrombectomy; Drug: 4°C saline infusion
- Mechanical thrombectomy combined with normothermic saline infusion (normothermia) group (Active Comparator): Patients received a total of 350 ml of roomtemperature saline infusion in addition to mechanical thrombectomy (MT).
  Interventions: Procedure: Mechanical thrombectomy; Drug: Normothermic saline infusion

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Mechanical thrombectomy
Drug: 4°C saline infusion — Patients received a total of 350 ml of 4°C saline infusion in addition to mechanical thrombectomy (MT).
  Arms: Mechanical thrombectomy combined with intra-arterial selective cooling infusion (hypothermia) group
Drug: Normothermic saline infusion — Patients received a total of 350 ml of roomtemperature saline infusion in addition to mechanical thrombectomy (MT).
  Arms: Mechanical thrombectomy combined with normothermic saline infusion (normothermia) group

SUMMARY:
A multicenter, prospective, open-label, blinded-endpoint, randomized controlled trial to assess the effectiveness and safety of catheter-based focal intracranial hypothermia combined with endovascular reperfusion therapy for patients with acute anterior circulation large artery occlusion.

DETAILED DESCRIPTION:
This trial aims to assess the effectiveness and safety of catheter-based focal intracranial hypothermia combined with endovascular reperfusion therapy for patients with acute anterior circulation large artery occlusion. This study used a stratified randomization method, with participants randomly allocated in a 1:1 ratio by a central network randomization system to either the mechanical thrombectomy (MT) combined with arterial selective cooling infusion (intravenous recombinant tissue plasminogen activator) (hypothermia) group or the MT combined with normal saline infusion (normothermia) group (hereinafter referred to as the hypothermia group or normothermia group). Randomization was stratified by ASPECTS score (≥8 or <8) and age (≥75 years or <75 years).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤85 years old.
2. Symptoms of sudden focal or general neurological impairment.
3. There may be a causal relationship between vascular occlusion and nerve function defect.
4. Time from symptom onset to randomization ≤24h.
5. The National Institutes of Health Stroke Scale (NIHSS) score was ≥6 points before randomization.
6. According to the judgment of the clinician, the operation path is reasonable, and the operation and operation related instruments can reach the disease smoothly.
7. Patients or their guardians can understand the purpose of the trial, voluntarily participate and sign a written informed consent, and are capable of receiving clinical follow-up.
8. Prior to randomization, CTA, MRA, or DSA confirmed the presence of anterior circulatory large vessel occlusion (internal carotid artery or M1segment).
9. The symptoms are aggravated by recurrent cerebral infarction in the same drainage basin and/or the pathogenesis is caused by decreased blood perfusion.

Exclusion Criteria:

1. Pre stroke mRS>1 score.
2. There are acute infarcts in both cerebral hemispheres and/or anterior and posterior circulation.
3. NIHSS≤6 points.
4. Cerebral hemorrhage/subarachnoid hemorrhage was confirmed by CT or MRI. 5.The presence of active bleeding, severe anemia, coagulation dysfunction, or an uncorrected bleeding tendency (Presence of at least one of the following laboratory tests: hemoglobin < 10g /dl, platelet count < 100,000 /μl, uncorrected INR>1.5, PT> 1 minute above the upper limit of normal, or heparin-related thrombocytopenia).

6.Patients with heart function of grade 1 or above, or with a clear history of acute or chronic heart dysfunction, are at greater risk of acute heart failure or fluid perfusion intolerance as determined by clinicians.

7. Severe heart, liver, kidney disease. 8.With malignant diseases such as malignant tumors, the expected survival time is less than 3 months.

9.Participating in other clinical trials, in the investigational phase or in the follow-up phase.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-2 at 90 days. | 90 days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-1 at 90 days | 90 days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Successful reperfusion rate | At the end of the operation
  Successful reperfusion was indicated by modified Thrombolysis in Cerebral Infarction (mTICI) grade 2b or 3.
Cerebral infarction volume was measured by CT or magnetic resonance DWI 72 hours to 7 days after operation | 72 hours to 7 days after procedure
  Cerebral infarction volume was measured by CT or DWI 72 hours to 7 days after operation.
Incidence of early neurological deterioration | Within 24 hours after procedure
  Early neurological deterioration was defined as an increase of 4 or more points on the NIHSS within 24 hours that was not attributable to intracerebral hemorrhage.
Rate of recurrent occlusion on MRA or CTA (postoperative 24 Hours to 7 Days) | postoperative 24 Hours to 7 Days
  Recurrent occlusion was measured by MRA or CTA 24 hours to 7 days after operation.

OTHER OUTCOMES:
Rate of symptomatic intracranial hemorrhage within 72 hours (Heidelberg Bleeding Classification) | Within 72 hours after procedure
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 72 hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma. The sICH was defined as ICH associated with a worsening of 4 or more points on the NIHSS or resulting in death, and cerebral herniation, which were not present at baseline.
Rate of coagulation disorders | 7 days
  Rate of coagulation disorders within 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China